CLINICAL TRIAL: NCT07288528
Title: A 2x2 Factorial, Randomized, Open-label Trial to Evaluate Neuromodulators and Cough Control Therapy in Patients With Refractory or Unexplained Chronic Cough (FORTITUDE)
Brief Title: A 2x2 Factorial, Randomized, Open-label Trial to Evaluate Neuromodulators and Cough Control Therapy in Patients With Refractory or Unexplained Chronic Cough
Acronym: FORTITUDE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FORTITUDE-01
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cough; Refractory Chronic Cough; Unexplained Chronic Cough; Cough Hypersensitivity Syndrome; Chronic Cough
Keywords: Cough; Chronic Cough; Morphine; Pregabalin; Non-Pharmacologic Therapy; Refractory Chronic Cough; Unexplained Chronic Cough
MeSH Terms: conditions — Cough; Chronic Cough; cough hypersensitivity syndrome | interventions — Morphine; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Morphine Sulphate (Experimental): Oral morphine sulphate given up to 5 mg twice daily.
  Interventions: Drug: Morphine Sulphate
- Morphine Sulphate + Cough Control Therapy (Experimental): Oral morphine sulphate given up to 5 mg twice daily and cough control therapy (5 virtual sessions delivered over 6 weeks by a trained physiotherapist and speech-language pathologist).
  Interventions: Combination Product: Morphine Sulphate + Cough Control Therapy
- Pregabalin (Experimental): Oral pregabalin given up to a maximum tolerated dose of 150 mg twice daily.
  Interventions: Drug: Pregabalin
- Pregabalin + Cough Control Therapy (Experimental): Oral pregabalin given up to a maximum tolerated dose of 150 mg twice daily and cough control therapy (5 virtual sessions delivered over 6 weeks by a trained physiotherapist and speech-language pathologist).
  Interventions: Combination Product: Pregabalin + Cough Control Therapy

INTERVENTIONS:
Drug: Morphine Sulphate — Oral morphine sulphate given up to 5 mg twice daily.
  Arms: Morphine Sulphate
Combination Product: Morphine Sulphate + Cough Control Therapy — Oral morphine sulphate given up to 5 mg twice daily and cough control therapy (5 virtual sessions delivered over 6 weeks by a trained physiotherapist and speech-language pathologist).
  Arms: Morphine Sulphate + Cough Control Therapy
Drug: Pregabalin — Oral pregabalin given up to a maximum tolerated dose of 150 mg twice daily.
  Arms: Pregabalin
Combination Product: Pregabalin + Cough Control Therapy — Oral pregabalin given up to a maximum tolerated dose of 150 mg twice daily and cough control therapy (5 virtual sessions delivered over 6 weeks by a trained physiotherapist and speech-language pathologist).
  Arms: Pregabalin + Cough Control Therapy

SUMMARY:
The FORTITUDE trial will provide head-to-head evidence on the benefits and harms of two commonly prescribed neuromodulators (low-dose morphine and pregabalin), the effectiveness of a virtual cough control therapy, exploratory assessment of potential synergy in combining these interventions, and the long-term outcomes of these treatments in patients with refractory or unexplained chronic cough.

DETAILED DESCRIPTION:
FORTITUDE (FactOrial Randomized TrIal To evalUate neuromoDulators and cough control thErapy) is a 6-week, 2x2 factorial, randomized, open-label trial with an extension observational phase up to 1 year. The trial will include Canadian hospital sites enrolling 124 patients. Patients ≥18 years old with either refractory or unexplained chronic cough will undergo 1:1:1:1 randomization to receive either low-dose morphine (up to 5 mg twice daily) or pregabalin (up to a maximum tolerated dose of 150 mg twice daily) with or without cough control therapy. The cough control therapy will consist of five virtual sessions delivered over 6 weeks by a trained physiotherapist and speech-language pathologist. Change from baseline in 24-hour cough frequency at 6 weeks represents the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years old) with either:
2. Refractory chronic cough (RCC), defined as having one or more identifiable causes of cough (asthma, allergic rhinitis, and/or GERD), but with previous trials of treatment targeting the underlying condition leading to no cough resolution; OR
3. Unexplained chronic cough (UCC), defined as having a cough lasting >8 weeks with (i) a normal chest X-ray/CT in the last 5 years and since the onset of chronic cough; (ii) FEV1 and FVC ≥80% predicted or >lower limit of normal (LLN); (iii) FEV1/FVC ≥0.7 or >LLN; (iv) no evidence of asthma; and (vi) no regular symptoms of nasal/reflux disease.

Exclusion Criteria:

1. Those who, in the opinion of the investigator, have previously tried low-dose morphine, pregabalin, and/or CCT with full intervention fidelity for the treatment of RCC/UCC;
2. Are currently taking morphine or pregabalin for the treatment of any indication (i.e., RCC/UCC or chronic pain);*
3. Are currently taking other centrally-acting medication (i.e., gabapentin, amitriptyline, dextromethorphan) for the treatment of any indication (i.e., RCC/UCC, seizures, or depression);*
4. Have a history of opioid or substance abuse that, in the opinion of the investigator, may interfere with the conduct of the study;
5. Are a current smoker, or ex-smoker with a >20 pack-year history who have abstained from smoking for <6 months;
6. Have cough due to angiotensin-converting enzyme inhibitor use;
7. Have symptoms of an upper respiratory infection within the last month that have not resolved;
8. Had an asthma exacerbation within the last month that requires an increase or start of an oral corticosteroid;
9. Have other primary pulmonary disorders, including pulmonary embolism, pulmonary hypertension, lung cancer, cystic fibrosis, radiologically-proven emphysema, interstitial lung disease, or severe bronchiectasis;
10. Have language, memory, cognitive, or psychiatric issues that may prevent optimal participation;
11. Have creatinine clearance <15 mL/min, including individuals with end-stage renal disease who require hemodialysis or peritoneal dialysis;
12. Have any other condition that, in the opinion of the qualified investigator, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant;
13. Have participated in another clinical trial of an investigational medicinal product within 30 days;
14. Pregnant or breastfeeding; or
15. Females of child-bearing potential who:

    1. Do not agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of 3 months.
    2. Acceptable methods of birth control include oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormone implant, double-barrier method, intrauterine devices, non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s), vasectomy of partner at least 6 months prior to screening.
    3. Females who are not of child-bearing potential will be defined as females who have undergone a sterilization procedure (e.g., hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening.

       * Participants taking any of the above medications at baseline will only be eligible if they are willing and medically able to safely discontinue them at least 2 weeks prior to the first study visit. Eligibility will be confirmed by the local study investigator prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24-hour cough frequency (coughs/hour) measured by the VitaloJAK ambulatory cough monitor at 6 weeks | 6 weeks

SECONDARY OUTCOMES:
Change from baseline in awake cough frequency (coughs/hour) measured by the VitaloJAK ambulatory cough monitor at 6 weeks | 6 weeks
Change from baseline in sleep cough frequency (coughs/hour) measured by the VitaloJAK ambulatory cough monitor at 6 weeks | 6 weeks
Change from baseline in cough bouts (defined by inter-cough intervals) measured by the VitaloJAK ambulatory cough monitor at 6 weeks | 6 weeks
Change from baseline in cough severity on the McMaster Cough Severity Questionnaire at 6 weeks | 6 weeks
Change from baseline in cough severity on the 100-mm visual analogue scale at 6 weeks | 6 weeks
Change from baseline in cough-specific quality of life on the Leicester Cough Questionnaire at 6 weeks | 6 weeks
Change from week 6 (end of randomized phase) in cough severity on the McMaster Cough Severity Questionnaire at 6 and 12 months | 6 and 12 months
Change from week 6 (end of randomized phase) in cough severity on the 100-mm visual analogue scale at 6 and 12 months | 6 and 12 months
Change from week 6 (end of randomized phase) in cough-specific quality of life on the Leicester Cough Questionnaire at 6 and 12 months | 6 and 12 months

OTHER OUTCOMES:
Proportion of patients with any adverse event for each intervention at 6 weeks, 6 months, and 12 months | 6 weeks, 6 months, and 12 months
Proportion of patients with treatment-related adverse events for each intervention at 6 weeks, 6 months, and 12 months | 6 weeks, 6 months, and 12 months
Proportion of patients with serious adverse events for each intervention at 6 weeks, 6 months, and 12 months | 6 weeks, 6 months, and 12 months
Proportion of patients with adverse events leading to treatment discontinuation for each intervention at 6 weeks, 6 months, and 12 months | 6 weeks, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Imran Satia, MD PhD, Principal Investigator — McMaster University; Wafa Hassan, MD, Study Chair — McMaster University; Elena Kum, Study Chair — McMaster University
Locations (5):
- Canada (5):
  - Respiratory Clinical Trials Centre, University of Calgary, Calgary, Alberta
  - Respiratory Research Lab, McMaster University, Hamilton, Ontario
  - St Joseph's Health Care London, London, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Quebec - University Laval, Québec, Quebec
  - Centre de recherche du Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec